CLINICAL TRIAL: NCT00873444
Title: Randomised, Controlled, Prospective, Multi-Centre, Post Market Surveillance Study Comparing a Ceramic-on-Metal Bearing and a Metal-on-Metal Bearing in Subjects Requiring Primary Total Hip Arthroplasty for Non-Inflammatory Degenerative Joint Disease
Brief Title: A Randomised Study to Compare Metal Ion Release and Long-term Performance of the Pinnacle™ Cup With a Ceramic-on-Metal or a Metal-on-Metal Bearing
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study progress very slow therefore terminated as other projects underway to investigate the same research question which will deliver results earlier
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT00/37
Record Dates: First submitted 2009-03-19; First posted 2009-04-01 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis; Post-traumatic Arthritis; Collagen Disorders; Avascular Necrosis; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis
Keywords: Hip; Cementless; Ceramic-on-Metal; Metal-on-Metal
MeSH Terms: conditions — Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1) Ceramic-on-Metal Bearing (Active Comparator): A cementless acetabular cup with ceramic liner for use in total hip replacement
  Interventions: Device: Pinnacle™ Acetabular System
- 2) Metal-on-Metal Bearing (Active Comparator): A cementless acetabular cup with metal liner for use in total hip replacement
  Interventions: Device: Pinnacle™ Acetabular System

INTERVENTIONS:
Device: Pinnacle™ Acetabular System — A cementless acetabular cup with ceramic liner for use in total hip replacement
  Arms: 1) Ceramic-on-Metal Bearing
Device: Pinnacle™ Acetabular System — A cementless acetabular cup with metal liner for use in total hip replacement
  Arms: 2) Metal-on-Metal Bearing

SUMMARY:
The purpose of this study is to monitor the performance and compare the metal ion release of two bearing combinations, ceramic-on-metal and metal-on-metal in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be randomly allocated to one of the bearing combinations and will be evaluated at regular intervals using, patient, clinical and x-ray assessments. Patients will also have blood samples taken at regular intervals to allow the metal ion levels to be determined.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature male or female subjects, aged between 20 and 75 years inclusive at the time of surgery.
* Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
* Subjects who, in the opinion of the Investigator, are able to understand this investigation co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects undergoing unilateral primary total hip replacement who are suitable for a cementless acetabular component and whose femoral and acetabular bone stock is suitable to receive implants, without the requirement for a bone graft.
* Subjects with radiographic evidence and primary diagnosis of non-inflammatory degenerative joint disease (NIDJD).
* Subjects with a pre-operative Harris Hip Score of less than or equal to 70 and a pain rating of at least moderate for the operative hip.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition, such as active infections, highly communicable diseases, neurological or musculoskeletal disorders that might affect weight-bearing and metastatic or neoplastic disease, that would compromise their participation and follow-up in this study.
* Subjects who currently have other metallic foreign bodies including trauma products and joint arthroplasties, unless known to be titanium alloy only.
* Patients who have received a total hip arthroplasty in the contralateral hip within the previous 12 months unless known to be titanium alloy only.
* Subjects who have undergone previous hip surgery on the operative hip (including previous hip/surface replacements, resection arthroplasty or surgical fusion of the hip).
* Subjects requiring a simultaneous bilateral hip operation.
* Subjects who, in the opinion of the investigator, will possibly require a separate joint replacement operation within the next two years, including revision operations.
* Subjects with an acute femoral neck fracture of the operative hip.
* Subjects who have undergone above knee amputation of the contralateral and/or ipsilateral leg.
* Subjects with compromised renal function.
* Subjects with a known allergy to metal (eg, jewellery).
* Subjects with an occupational exposure to cobalt, chromium, molybdenum, titanium or nickel.
* Subjects who have ingested medication or vitamins containing cobalt, chromium, molybdenum, titanium or nickel within the last 12 months, or intend to ingest such substances over the next 2 years.
* Subjects who have undergone systemic steroid therapy, excluding inhalers, in the three months prior to surgery.
* Women who are pregnant.
* Subjects who are prisoners, known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical study with an investigational product in the last 12 months.
* Subjects who are currently involved in any injury litigation claims.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Cobalt metal ion levels in the blood at 2 years post surgery | 2 years post-surgery

SECONDARY OUTCOMES:
Kaplan-Meier survivorship calculations | Annually
Oxford Hip Score | 6 weeks, 6 months, and Annually
UCLA Score | 6 weeks, 6 months, and Annually
Pain Visual Analogue Scale | 6 weeks, 6 months, and Annually
Harris Hip Score | 6mths, 1yr, 2yrs, 5yrs and 10yrs post-surgery
Radiographic analysis | 6 weeks, 6mths, 1yr, 2yrs, 5yrs and 10yrs post-surgery
Blood metal ion levels | pre-discharge, 6 weeks, 6mths, 1yr, 2yrs, 5yrs and 10yrs post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Garmisch-Partenkirchen, Garmisch-Partenkirchen, Germany